CLINICAL TRIAL: NCT00829140
Title: A 56-Day , Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Effect of Lorcaserin Hydrochloride on Energy Metabolism and Food Intake in Overweight and Obese Patients (TULIP)
Brief Title: To Assess the Effect of Lorcaserin Hydrochloride on Energy Metabolism and Food Intake
Acronym: TULIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: APD356-014
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2010-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — lorcaserin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo
- Lorcaserin 10mg BID (Experimental)
  Interventions: Drug: Lorcaserin 10mg BID

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo BID
Drug: Lorcaserin 10mg BID
  Arms: Lorcaserin 10mg BID

SUMMARY:
The purpose of this study is to evaluate the effect of lorcaserin on energy metabolism and food intake in obese and overweight patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged between 18 and 65 years (inclusive)
2. Body Mass Index (BMI) is 27.0 to 45.0 kg/m2, inclusive
3. Able to give signed informed consent
4. Ambulatory and able to perform exercise program (Arena Healthy Lifestyle Program, see Appendix 1)
5. Eligible male and female patients must agree not to participate in a conception process
6. Considered to be in stable health in the opinion of the Investigator

Exclusion Criteria:

1. Prior participation in any study of lorcaserin.
2. Participants who are current smokers or have smoked within the previous 6 months. No smoking will be allowed during the study.
3. Clinically significant new illness in the 1 month before screening
4. Not suitable to participate in the study in the opinion of the Investigator including an existing physical or mental condition that prevents compliance with the protocol
5. Recent history (within 6 months before entering the study) of major depression, anxiety, or other psychiatric disease requiring treatment with prescription medication. SSRI's, SNRI's, and other medications must meet washout requirements.
6. Significant dislike or allergy to foods used during the food intake tests
7. History of any of the following cardiovascular conditions:

   * Myocardial infarction (diagnosed by cardiac enzyme[s] and/or diagnostic ECG), CVA, TIA or RIND within 3 months of screening; cardiac arrhythmia requiring medical or surgical treatment within 3 months of screening
   * Unstable angina
   * History of congestive heart failure caused by insufficiency, damage, or stenosis of any heart valve
   * History of pulmonary artery hypertension
8. Positive result of HIV, hepatitis B or hepatitis C screens
9. Recent treatment (i.e., within 1 month of the screening visit) with over-the-counter weight loss products or appetite suppressants (including herbal weight loss agents), or within 3 months with a prescription anti-obesity drug (e.g., phentermine, sibutramine, orlistat)
10. Participated in any clinical study with an investigational drug, biologic, or device within 1 month prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To assess the effect of lorcaserin on 24h energy metabolism (measured in a respiratory chamber) after 56 days of treatment.

SECONDARY OUTCOMES:
To assess the ongoing safety of lorcaserin

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151
- [Derived] Martin CK, Redman LM, Zhang J, Sanchez M, Anderson CM, Smith SR, Ravussin E. Lorcaserin, a 5-HT(2C) receptor agonist, reduces body weight by decreasing energy intake without influencing energy expenditure. J Clin Endocrinol Metab. 2011 Mar;96(3):837-45. doi: 10.1210/jc.2010-1848. Epub 2010 Dec 29. PMID 21190985